CLINICAL TRIAL: NCT07135440
Title: The Association of Biomarkers Detected by Optical Coherence Tomography Angiography (OCTA) of the Macula With Cognitive Functions in Patients With Type 2 Diabetes
Brief Title: The Potential of Optical Coherence Tomography Angiography (OCTA) to Detect Early Cognitive Dysfunction in Diabetic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. Sefic Eye Polylcinic and Optical Studio (Other)
Responsible Party: Principal Investigator, Aida Pidro Gadzo, General hospital "prim.dr.Abudlah Nakas" and Dr. Sefic Eye Polyclinic and Optical Studio, Dr. Sefic Eye Polylcinic and Optical Studio
Other Study IDs: OCTA-DM2-Cognition-01
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus Diabetic Retinopathy Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Group I: Patients with type 2 diabetes without clinically detectable diabetic retinopathy changes
  Interventions: Device: OCT angiography RTVue XR Avanti; Optovue, Inc, Fremont, California, USA
- Group II: Patients with type 2 diabetes with non-proliferative diabetic retinopathy
  Interventions: Device: OCT angiography RTVue XR Avanti; Optovue, Inc, Fremont, California, USA
- Group III: Healthy individuals (control group), age and gender mached
  Interventions: Device: OCT angiography RTVue XR Avanti; Optovue, Inc, Fremont, California, USA

INTERVENTIONS:
Device: OCT angiography RTVue XR Avanti; Optovue, Inc, Fremont, California, USA — OCTA is a fast, non-invasive, and contactless imaging technique that enables detailed visualization of the retinal microvasculature by tracking erythrocyte movement within blood vessels in real time. It provides layer-by-layer analysis of the retina and choroid without the need for intravenous contrast, significantly reducing patient risk and improving accessibility. Increasing evidence suggests that neurodegenerative and vascular changes precede clinically visible signs of disease, making OCTA a valuable diagnostic tool for early detection of diabetic retinopathy before it can be confirmed through standard fundus examination. The MoCA test includes assessments of executive functions, high-level language abilities, and complex visuospatial tasks, making it suitable for detecting even mild cognitive dysfunction.
  Other Names: MoCA scale for cognitive assesment

SUMMARY:
Diabetic Retinopathy (DR) is one of the most common complications of diabetes, and its association with cognitive dysfunctions is becoming an increasingly frequent research interest. Non-proliferative diabetic retinopathy (NPDR) encompasses early changes at the microvascular level, which can be detected quantitatively and qualitatively through optical coherence tomography angiography (OCTA) well before the first symptoms of this disease appear. Cognitive dysfunction is often unrecognized in the early stages of diabetes. This research will focus on examining the association between OCTA parameters and cognitive functions in patients with NPDR. The aim of this study is to investigate the correlation between OCTA parameters and cognitive functions in patients with NPDR using the Montreal Cognitive Assessment (MoCA) scale to assess cognitive abilities and to establish a connection between OCTA biomarkers and changes in cognitive function. Patients with type 2 diabetes will be included in the study. Patients with proliferations and diabetic macular edema affecting the center and reducing visual acuity will be excluded to minimize error in cognitive function assessment caused by vision impairment. OCTA will be used to analyze microvascular changes in the retina, including capillary density and areas of the avascular zone. At the same time, the MoCA scale will be used to assess cognitive function, focusing on aspects of memory, attention, executive function, and orientation. Data analysis will investigate correlations between OCTA parameters, the presence of diabetic retinopathy-related changes in the eye fundus, as well as the stage of retinopathy and MoCA scale scores, taking into account factors such as diabetes duration, previous diabetes treatment, lipid status, anthropometric parameters, and glycemic control. The results of this research are expected to provide better insight into the early diagnosis of cognitive dysfunctions in patients with diabetes, thereby contributing to the development of targeted interventions.

DETAILED DESCRIPTION:
OCTA represents a potential alternative for early detection of vascular abnormalities. OCTA algorithms generate an image, most commonly sized 3x3 mm or 6x6 mm, which is conventionally segmented into four zones: superficial retinal plexus, deep retinal plexus, outer retina, and choriocapillaris. OCTA enables monitoring of retinal vascular changes over time and allows early detection of microcirculatory abnormalities.

Cognition is the process by which the human brain receives information from the external environment, processes it, and transforms it into internal psychological activities for acquiring or applying knowledge. It includes memory, language, visuospatial skills, executive function, calculation, comprehension, and judgment. Various cognitive function tests have been developed through years of research. The most commonly used screening test for general cognitive function is the Mini-Mental State Examination (MMSE), while a more recent and sensitive tool is the Montreal Cognitive Assessment (MoCA). The MoCA test includes assessments of executive functions, high-level language abilities, and complex visuospatial tasks, making it suitable for detecting even mild cognitive dysfunction. Although these tests can assess a patient's cognitive level, they cannot confirm the presence of cerebral microvascular disease.

Numerous studies suggest a link between diabetes mellitus and cognitive impairment. While cognitive decline is not specific to diabetes, it is now recognized as a complication of the disease. In studies involving older populations, patients with diabetes demonstrated a higher risk of developing Alzheimer's disease and other forms of dementia. Since diabetes affects the entire vascular system, it is assumed that changes in the retinal microvasculature may reflect the general vascular condition of the body, including changes in the brain. Studies have shown that patients with advanced stages of DR often exhibit reduced cerebral blood flow, further contributing to cognitive decline.

Research also suggests that early interventional treatments, such as improved glycemic control and therapies aimed at enhancing vascular function, could reduce the risk of cognitive deterioration. There is growing evidence that changes in the retinal microvascular structure may reflect similar alterations in cerebral vascular structures, given that the retina and brain share common embryological and anatomical characteristics.

This study differs from previous ones as it focuses exclusively on the early stages of NPDR, including patients with diabetes who show no detectable changes on fundoscopy. This minimizes the risk of errors on the MoCA scale, since patients with reduced visual acuity due to macular edema or proliferative changes may score falsely low, leading to inaccurate assessments of their cognitive function.

Moreover, the MoCA scale used in this study is more comprehensive, providing a detailed evaluation of cognitive function, unlike previous studies which often used shorter tests or focused on isolated cognitive domains. The results of this research will define the specific OCTA parameters associated with cognitive function, making them potential biomarkers for detecting both ophthalmological and neurological disorders in diabetic patients.

Aim

1. To examine whether changes detected in the retinal layers and retinal vasculature using OCTA correlate with cognitive impairment in patients with type 2 diabetes.
2. To investigate whether the decline in cognitive function is more pronounced in patients with more advanced stages of the disease.
3. To identify retinal microvascular biomarkers using OCTA that could be used for the early detection of cognitive impairment and the severity of diabetic retinopathy in affected patients.

Working hypothesis:

Patients with diabetic retinopathy exhibit reduced cognitive function compared to patients without diabetic retinopathy. An increase in macular ischemia leads to a decline in cognitive function.

A prospective cross-sectional clinical study will be conducted at the General Hospital "Prim. Dr. Abdulah Nakaš" and the private ophthalmology clinic "Dr. Sefić" in Sarajevo, from January 1, 2025, to January 1, 2026, or until the target number of participants is reached. Approval from the Ethics Committee for conducting the study was obtained on January 9, 2025 (Reference No. 26-213-114/25). A total of 210 participants will be included in the study, who will be divided into three groups of 70 based on clinical, laboratory, and ophthalmological indicators:

* Group A: Patients with type 2 diabetes without diabetic retinopathy (DR) changes,
* Group B: Patients with type 2 diabetes with non-proliferative diabetic retinopathy (NPDR),
* Group C: Healthy individuals (control group). Basic anamnesis data will be collected for all participants using a specially designed form. The form will include basic demographic data (name and surname, age, gender), disease duration, presence of comorbidities, current treatment methods, and information on smoking and alcohol consumption. Laboratory parameters will be used for each participant, not older than one month, including: plasma glucose concentration (FPG), HbA1c, lipid profile, renal function parameters (urea and creatinine), and systolic and diastolic blood pressure.

Each participant will be fully informed about the study and allowed to ask additional questions. Participation will be confirmed by signing an informed consent form, which clearly outlines the study details. The study will adhere to the principles of the Nuremberg Code, the latest revision of the Declaration of Helsinki, the Law on Health Protection ("Official Gazette of the Federation of Bosnia and Herzegovina," No. 46/10), and the Law on the Rights, Duties, and Responsibilities of Patients ("Official Gazette of the Federation of Bosnia and Herzegovina," No. 40/10). Data will be collected in accordance with ethical principles, ensuring participant privacy and data confidentiality. The data obtained will be used solely for this research. Ethical approval was requested from the Ethics Committee of the General Hospital "Prim. Dr. Abdulah Nakaš" in Sarajevo.

Participants will first complete the MoCA test, version 7.1, translated into Croatian. The MoCA test is a widely used screening tool for detecting mild cognitive impairment and early signs of dementia. It can help identify individuals at risk for Alzheimer's disease and screen for conditions such as Parkinson's disease or the effects of brain tumors. MoCA is a simple tool that quickly assesses cognitive impairment, including the ability to understand, reason, and remember.

The test consists of 14 different tasks with a maximum total score of 30 points. During the test, patients will be given instructions for each task, with an explanation of the test duration and purpose. The test lasts 10-12 minutes and assesses seven areas of cognitive function:

1. Visuospatial/executive function - the participant connects alternating numbers and letters, draws a three-dimensional cube, and draws a clock showing 4:05 (3 tasks, 5 points total);
2. Naming - the participant is shown images of three animals and asked to name them (1 point each, 3 points total);
3. Attention - includes four tasks: repeating numbers forward and backward, identifying the letter "A" in a sequence, and subtracting 7 from 100 backward (6 points total);
4. Language - repeating two sentences exactly as spoken and listing as many words as possible beginning with the letter T within one minute (3 points total);
5. Abstract thinking - identifying common features between two concepts, after a similar example is provided (2 points total);
6. Delayed recall - remembering and recalling five words that were given at the beginning of the test after five minutes (5 points total);
7. Orientation - answering questions about the date, month, year, day of the week, city, and place where the person is located (6 points total).

The total possible score is 30 points. If a person has 12 or fewer years of formal education, 1 point is added to the total score. After completing the test, the total score and individual section scores will be calculated for each participant.

Test results are interpreted as follows:

1. Normal cognition: 26-30 points
2. Mild cognitive impairment: 18-25 points
3. Moderate impairment: 10-17 points
4. Severe impairment: <10 points

The ophthalmological examination will include:

1. Determination of best corrected visual acuity,
2. Measurement of intraocular pressure using Goldmann applanation tonometry,
3. Slit-lamp examination of the anterior segment,
4. Slit-lamp examination of the posterior segment with detailed notation of microaneurysms, dot and blot hemorrhages, cotton wool spots, and hard exudates,
5. OCTA (Optical Coherence Tomography Angiography) with qualitative and quantitative biomarker analysis.

OCTA is a fast, non-invasive, and contactless imaging technique that enables detailed visualization of the retinal microvasculature by tracking erythrocyte movement within blood vessels in real time. It provides layer-by-layer analysis of the retina and choroid without the need for intravenous contrast, significantly reducing patient risk and improving accessibility. Increasing evidence suggests that neurodegenerative and vascular changes precede clinically visible signs of disease, making OCTA a valuable diagnostic tool for early detection of diabetic retinopathy before it can be confirmed through standard fundus examination. The OCTA device used will be the RTVue XR Avanti (Optovue, Inc., Fremont, California, USA).

The following quantitative OCTA biomarkers will be considered:

1. Size and perimeter of the foveal avascular zone (FAZ) - FAZ is the central avascular area of the macula, and its size increases with DR progression, indicating retinal ischemia. FAZ perimeter measures the length of the avascular zone border; a larger perimeter is associated with worsening ischemia and DR progression.
2. Vessel density - refers to the percentage of retinal area filled with vessels; it decreases as DR progresses, indicating microvascular network loss.
3. Perfusion density - indicates the volume of blood circulating through retinal capillaries; a decrease may signal early vascular abnormalities in diabetes.
4. Number of parafoveal capillary dropouts - represents areas of capillary loss or ischemia in the parafoveal region; an increased number indicates advancing microangiopathy.
5. Perifoveal area (PeriFAZ) - the vascular network surrounding the FAZ; reduced perfusion density in this area suggests early ischemic damage in diabetic retinopathy.
6. Fractal dimension (FD) - a mathematical parameter describing the complexity of the retinal vascular network; reduced FD values are associated with capillary structure loss in DR.

The expected scientific contribution of this research is the identification of an early correlation between retinal microvascular changes and cognitive decline in patients with type 2 diabetes. It is anticipated that these changes will be more pronounced in eyes showing signs of non-proliferative diabetic retinopathy, especially in its advanced stages. Such findings could enable timely ophthalmologic and neurologic interventions, thereby improving the quality of life for individuals with diabetes.

One of the key objectives of the study is to confirm the hypothesis that OCTA can serve as a non-invasive, quantitative biomarker for the early detection of cerebral vascular changes, reflected through microvascular alterations in the retina. In this way, OCTA could be positioned as a valuable tool for early identification of cognitive changes-potentially even before the appearance of classical neurological symptoms or findings on radiological imaging.

This research opens a new perspective in understanding the connection between ocular and cerebral vascular health and lays the foundation for future care models for diabetic patients, based on a multidisciplinary approach and early detection of the risk for cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* diagnosed type 2 diabetes mellitus
* literacy, transparent optical media, and visual acuity sufficient to independently complete tasks on the Montreal Cognitive Assesment scale (MoCA) scale (>0.5),
* signed informed consent form allowing participation in the study and use of the data for research and educational purposes.

Exclusion Criteria:

* illiteracy,
* lack of necessary test results,
* best corrected visual acuity less than 0.5,
* prior anti-VEGF treatment or pars plana vitrectomy (PPV),
* proliferative diabetic retinopathy (PDR),
* diabetic macular edema involving the center,
* non-transparent optical media,
* legal incompetence due to psychiatric disorders or intellectual disability,
* acute and chronic inflammatory conditions, and
* malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes mellitus, aged 18 years to 80 years, undergoing routine ophthalmologic examination at the General Hospital "Prim. Dr. Abdulah Nakaš" and "dr Sefic Eye Polyclinic and Optical Studio" in Sarajevo. Participants must have a confirmed diagnosis of diabetes mellitus type 2 and be able to complete the MoCA cognitive assessment.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative retinal microcirculation parameters detected on OCTA | Day 1
  Retinal vessel density will be assessed using Optical Coherence Tomography Angiography (OCTA), focusing on specific retinal layers such as the superficial and deep capillary plexus. Quantitative analysis will include vessel density (%) and foveal avascular zone (FAZ) parameters. These measurements aim to identify microvascular changes potentially associated with cognitive function in patients with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
MoCA Score for Cognitive Function Assessment | Day 1
  The Montreal Cognitive Assessment (MoCA) is a validated cognitive screening tool that assesses multiple cognitive domains, including memory, attention, language, abstraction, and orientation. The total score ranges from 0 to 30, with lower scores indicating greater cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- dr Sefic Eye Polyclinic and Optical Studio, Sarajevo, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No